CLINICAL TRIAL: NCT07285707
Title: Acupuncture for Long COVID - A Pragmatic Pilot Study
Brief Title: Acupuncture and Chinese Herbal Medicine for Long COVID
Acronym: ACUCM-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VINJ011; VINJ011 (Other: SCUHS)
Record Dates: First submitted 2025-11-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
Keywords: long covid; acupuncture for long COVID; Chinese medicine for long COVID; Chinese herbal medicine for long COVID; acupuncture; Chinese herbal medicine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pragmatic experimental arm (Experimental): Single-arm study looking at feasibility and acceptability of acupuncture treatment for 5 patients and acupuncture and Chinese herbal medicine for 5 patients
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — The investigators have developed a list of core acupoints, which will be used by all clinicians for each specific TCM diagnosis pattern identified in each patient. Similarly, a list of common herbal formulas, that we will keep in stock based on the specific diagnosis patterns, has been developed. Clinicians will have the option of using additional acupoints as necessary and will be asked to record and explain any variations from the core protocol.
  1. Residual Heat: LI-11, KI-6;Bai He Gu Jin Tang
  2. Residual Phlegm: ST-40, Sp-9;Ban Xia Bai Zhu Tian Ma Tang,Er Chen Tang
  3. Deficiency of Spleen: SP-3, ST-36;Gui Pi Tang,Xiang Sha Liu Jun Zi Tang
  4. Lung Qi Deficiency with Dampness: LU-9, LU-7;Zhi Sou San,Er Chen Tang
  5. Blood Stagnation: SP-10, SP-6;Xue Fu Zhu Yu Tang,Tao Hong Si Wu Tang
  6. Deficiency of Lung: LU-9, LU-7; Bu Fei Tang
  7. Liver Qi Stagnation: LV-3, PC-6;Xiao Yao San, Chai Hu Shu Gan Tang
  8. Yin Deficiency: KI-6, SP-6;Liu Wei Di Huang Wan
  9. Deficiency of Kidney: KI-3, KI-6;

SUMMARY:
List of the Hypothesis:

Primary hypothesis: A flexible acupuncture and Chinese herbal medicine protocol will be feasible, acceptable, and useful for the treatment of long COVID.

Secondary hypothesis: Long COVID patients receiving acupuncture treatment or acupuncture treatment and Chinese herbal supplements over an 8-week period will see improvements in their symptoms, function, and quality of life measurements.

Specific Aims of This Research (Purpose of the study):

To study the feasibility, acceptability and utility of an acupuncture and Chinese herbal supplement treatment protocol for patients with long COVID and preliminarily assess the effects of treatment.

Currently Available Research on This Subject:

Studies indicate that acupuncture can effectively treat symptoms that are similar to those often seen in long COVID patients. Additionally, recent studies and clinical evidence suggest that there is substantial potential for acupuncture in the treatment of long COVID. Acupuncture may be beneficial because it can address many symptoms simultaneously with a single intervention, whereas symptom clusters can be difficult to manage with pharmaceuticals due to the need for multiple pharmaceutical agents.

Summary of the research protocol/methodology:

Five patients will receive acupuncture treatment, and five patients will receive acupuncture and Chinese herbal medicine. Each participant will receive 16 acupuncture treatments over the course of eight weeks (i.e., twice per week). Each treatment session will last for 30 minutes. Follow-up will occur at 12 weeks (i.e., four weeks after the final treatment session).

Significance of this research to the health and welfare of general public:

There is currently not a single, specific treatment for long COVID. If acupuncture treatment alone and/or acupuncture and Chinese herbal medicine combined are feasible, acceptable, and efficacious in the improvement of long COVID symptoms, it will offer patients additional treatment options, which may help some patients to avoid pharmaceutical treatment side effects or polypharmacy challenges.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

  * We will include adults of any age in our study. Adults of all ages can experience long COVID symptoms, although it is more common in older adults

    • Confirmed and documented COVID-19 illness (confirmed by healthcare provider or test; acceptable documentation includes but is not limited to a doctor's note or a photo of test result)
  * COVID-19 illness is a necessary precursor to the development of long COVID

    • Experiencing at least one of the following common long COVID symptoms for at least 4 weeks after confirmed COVID-19 illness:
  * Fatigue or post-exertional malaise,
  * Dyspnea, cough,
  * Brain fog, sleep disturbance, depression, anxiety,
  * Arthralgia, myalgia, or
  * Constipation, diarrhea, stomach pain
* Over 200 different long COVID symptoms have been identified. The proposed study is a small pragmatic pilot study which only plans to enroll 10 participants. It is necessary to limit inclusion to some of the most common symptoms to ensure that the findings are broadly relevant across the long COVID patient population.

  * The symptoms were not present prior to the confirmed COVID-19 illness

    o If the symptoms were present prior to the confirmed COVID-19 illness, then they are most likely attributable to a cause other than long COVID
  * Willingness to comply with the treatment schedule

    o It is important that all those who qualify for the study are willing to comply with the protocol that is being adopted. If the patient is not willing to attend acupuncture treatment sessions or comply with the supplement schedule, then they may not be enrolled in the study.
  * Ability to read and understand English o Informed consent will be in the English language. Inability to read and understand English will interfere with provision of informed consent. Moreover, compliance is a potential issue with herbal supplementation. Recruiting patients who are able to read and understand English instructions for supplement intake will help to improve compliance with the protocol.
  * Ability to provide informed consent o It is important that participants are aware that they are required to provide written informed consent before they are allowed to participate. Some individuals who are eligible might be unwilling to sign the informed consent form.

Exclusion Criteria:

* • Under 18 years of age

  * Pulmonary fibrosis or on continuous oxygen treatment
  * Certain preexisting conditions:

    * Diagnosed with Alzheimer's or demonstrating onset of dementia
    * Uncontrolled hypertension, diabetes, or autoimmune conditions
    * Other comorbid conditions that might imitate long COVID symptoms
  * Undergoing cancer treatments
  * Use of acupuncture or Chinese medicine in the past three months
  * Involved in health-related litigation or legal claims
  * Missing either baseline visit and deemed unlikely to comply with the study protocol
  * Pregnant or breastfeeding or trying to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementing a Combined Acupuncture and Chinese Herbal Medicine Intervention for long COVID | From enrollment to the final follow-up at 12 weeks
  Feasibility will be measured through a feasibility assessment questionnaire which will evaluate recruitment, retention, and adherence metrics across the 12-week intervention and the final follow-up. Feasibility indicators will be summarized as proportions and descriptive statistics to evaluate the practicality of the study procedures and protocol implementation.

SECONDARY OUTCOMES:
Patient-Reported Acceptability of the Study Procedures and Treatments | Week 12 (final follow-up).
  Acceptability will be evaluated using a participant satisfaction questionnaire administered at the end of the 12-week intervention. The survey includes Likert-scale items (1 = very dissatisfied to 5 = very satisfied) assessing participants' comfort with study procedures, satisfaction with the acupuncture and herbal treatment, and willingness to recommend participation to others. Mean scores will be calculated; higher scores indicate greater acceptability and satisfaction with the study protocol and treatment experience
Clinician-Reported Acceptability of the Study Protocol | Week 12 (final follow-up).
  Clinician acceptability will be measured through a self-administered survey at the end of the 12-week intervention. The survey uses a 5-point Likert scale (1 = very dissatisfied to 5 = very satisfied) to assess satisfaction with the clinical feasibility, workflow, and perceived patient benefit of the combined acupuncture and herbal medicine protocol. Scores will be averaged, and higher scores indicate greater clinician-reported acceptability.
Change in Health-Related Quality of Life Measured by PROMIS-29 v2.1 | Baseline, Week 4, Week 8, and Week 12.
  Quality of life will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS-29 v2.1) at baseline, mid-intervention, and post-intervention. The PROMIS-29 measures physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and social participation. Each domain produces a standardized T-score (mean = 50, SD = 10). Higher scores represent better functioning for positive domains and greater symptom burden for negative domains. Changes from baseline to Week 12 will reflect improvements or declines in overall quality of life.
Change in Symptom Burden Measured by the Symptom Burden Questionnaire for Long COVID (SBQ™-LC) | Baseline, Week 8, and Week 12.
  Symptom burden will be assessed using the Symptom Burden Questionnaire for Long COVID (SBQ™-LC). At baseline, participants complete all domains; at Weeks 8 and 12, they complete up to four domains corresponding to their most bothersome baseline symptoms, as well as the mandatory Mental Health and Well-Being domain. Each item is rated from 0 (no symptom) to 10 (worst possible symptom). Higher scores indicate greater symptom severity. Domain and total scores will be compared across time points to evaluate changes in symptom burden.
Change in Whole Health Person Index (WHPI) | Baseline, Week 8, and Week 12.
  Overall well-being will be measured using the Whole Health Person Index (WHPI), a 0-100 scale that assesses physical, emotional, and social wellness. Higher scores indicate better overall health and life balance. The change in WHPI from baseline to Week 12 will be used to evaluate perceived improvements in general well-being associated with the intervention.
Change in Laboratory Biomarkers - Complete blood count | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes complete blood count (CBC) with differential. Changes in this marker will indicate biological trends in inflammation.
Incidence and Severity of Adverse Events Associated with Acupuncture and Herbal Medicine | Throughout the 12-week study period
  Safety will be monitored throughout the 12-week study by documenting adverse events (AEs) and serious adverse events (SAEs) related to acupuncture or herbal supplementation. Each event will be recorded in Qualtrics using the Adverse Event Form and graded as mild, moderate, or severe per Institutional Review Board (IRB) and Common Terminology Criteria for Adverse Events (CTCAE v5.0) guidelines. Frequency and type of AEs will be summarized descriptively as counts and percentages.
Change in Laboratory Biomarkers - Comprehensive metabolic panel | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes complete comprehensive metabolic panel (CMP). Changes in this marker will indicate biological trends in inflammation and metabolic function.
Change in Laboratory Biomarkers - C-reactive protein | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes C-reactive protein (CRP). Changes in this marker will indicate biological trends in inflammation.
Change in Laboratory Biomarkers - Erythrocyte sedimentation rate | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes erythrocyte sedimentation rate (ESR). Changes in this marker will indicate biological trends in inflammation.
Change in Laboratory Biomarkers - Tumor necrosis factor-alpha | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes tumor necrosis factor-alpha. Changes in this marker will indicate biological trends in inflammation and metabolic function.
Change in Laboratory Biomarkers - thyroid panel | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Test includes thyroid panel. Changes in this marker will indicate biological trends in metabolic function.
Change in Laboratory Biomarkers - Vitamin D levels. | Baseline and Week 8.
  Laboratory values will be compared from baseline to Week 8 to assess physiological effects of the intervention. Tests include vitamin D levels. Changes in these markers will indicate biological trends in inflammation and metabolic function.

CONTACTS AND LOCATIONS:
Locations (1):
- SCUHS, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: No